CLINICAL TRIAL: NCT02240563
Title: Long-term Follow-up After Treatment of Chronic Autoimmune Thyroiditis With Low Level Laser
Brief Title: Low Level Laser Therapy for Autoimmune Thyroiditis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Danilo Bianchini Hofling, MD, University of Sao Paulo General Hospital, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAPPesq 11459
Record Dates: First submitted 2014-06-23; First posted 2014-09-15 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Autoimmune Thyroiditis
Keywords: autoimmune thyroiditis; LLLT; safety; ultrasound
MeSH Terms: conditions — Thyroiditis, Autoimmune | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low-level laser therapy (Experimental): This group of patients was treated with a continuous wave diode laser device (830 nanometer, infrared) with a beam area of 0.002827 cm2 using the punctual method on the continuous emission mode at an output power of 50 milliwatts and a fluence of 707 Joules/cm2 six years before.
  Interventions: Procedure: Low-level laser therapy
- Non laser ordinary red light (Placebo Comparator): This group of patients was treated using the same method and equipment, except that a non laser ordinary red light, an output power of 0.1 Watt and a fluence of 1.41 Joules/cm2 and an irradiance value of 0.0002827 Watts/cm2 (the placebo), indistinguishable from the laser beam, was used. Therefore, the patients were blinded to which treatment they received.
  Interventions: Procedure: Non laser ordinary red light

INTERVENTIONS:
Procedure: Low-level laser therapy
  Other Names: Low-power laser therapy
  Arms: Low-level laser therapy
Procedure: Non laser ordinary red light
  Other Names: Placebo
  Arms: Non laser ordinary red light

SUMMARY:
INTRODUCTION: Chronic autoimmune thyroiditis (TCA) is the main cause of acquired hypothyroidism, which requires continuous treatment with levothyroxine (LT4). A randomized, placebo-controlled trial including 43 patients with hypothyroidism caused by TCA without nodules on ultrasonography study (US) was conducted from March 2006 to March 2009 (NCT01129492). Among them, 23 were submitted to low-level laser therapy (LLLT) and 20 to placebo. The LLLT was effective in improving the echogenicity, the volume and of the thyroid vascularization pattern by US. There was also improvement in the thyroid function and reduction of serum thyroid peroxidase antibodies (TPOAb). Although the results have shown promising and LLLT has shown to be safe in many study models, the long-term LLLT actions on the thyroid parenchyma are unknown. Thus, the objective of this study is to perform biochemical tests and thyroid US six years after the clinical trial interventions to evaluate levothyroxine dose, serum levels of autoantibodies and, especially, the frequency and nature of nodules in the gland and then compare these variables between LLLT and placebo groups. METHODS: This study will include the trial participants performed six years before. The levothyroxine dose and serum levels of thyrotropin (TSH), T3, T4, free T4, TPOAb and anti-thyroglobulin antibodies (TgAb) will be evaluated in these patients. The thyroid US will assess the texture (with particular attention to identifying nodules), echogenicity, volume, as well as vascularization of the gland. The US nodules features, such as dimensions, shape, margins, extracapsular invasion, echogenicity, texture, hypoechoic halo, calcification, internal content, vascularization pattern and resistivity index will be searched. Regional lymph nodes and other characteristics will be also investigated. The USs will be carried out by only one examiner who will be blinded for the previously performed intervention (LILT or placebo). The same investigator will execute a fine needle aspiration (FNA) of patients with thyroid nodules. The cytological analysis of the material collected from the nodules will be undertaken by a pathologist who will be also blinded for the treatment assignments. RESULTS: The following variables will be compared between the two groups: levothyroxine doses, antithyroid antibodies, US parameters, thyroid nodules (if detected) and in this case, the result of their respective FNA.

ELIGIBILITY:
Inclusion Criteria:

All patients who have hypothyroidism caused by autoimmune thyroiditis included in the randomized, placebo controlled clinical trial (NCT01129492)

-

Exclusion Criteria:

All patients who have hypothyroidism caused by autoimmune thyroiditis included in the aforementioned trial (NCT01129492) who underwent surgery and/or therapeutic administration of radioiodine for thyroid diseases during the period between the initial assessment of patients up to the present study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2014-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Thyroid Nodules as a Measure of Safety | Six Years after Each Patient Treatment

SECONDARY OUTCOMES:
Serum Levels of Anti-Thyroglobulin Antibodies as a Measure of Long Term Efficacy | Six Years after Each Patient Treatment

OTHER OUTCOMES:
The Levothyroxine Required Dose as a Measure of Long-Term Efficacy | Six Years after Each Patient Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cristina Chammas, MD, Study Director — University of Sao Paulo General Hospital; Carlos Alberto Buchpiguel, PhD, Study Chair — University of Sao Paulo General Hospital; Danilo B Höfling, MD, Principal Investigator — University of Sao Paulo General Hospital
Locations (2):
- Brazil (2):
  - University of Sao Paulo General Hospital, Radiology Institute, São Paulo
  - University of Sao Paulo General Hospital, São Paulo

REFERENCES:
- [Background] Hofling DB, Chavantes MC, Juliano AG, Cerri GG, Knobel M, Yoshimura EM, Chammas MC. Low-level laser in the treatment of patients with hypothyroidism induced by chronic autoimmune thyroiditis: a randomized, placebo-controlled clinical trial. Lasers Med Sci. 2013 May;28(3):743-53. doi: 10.1007/s10103-012-1129-9. Epub 2012 Jun 21. PMID 22718472
- [Background] Hofling DB, Chavantes MC, Juliano AG, Cerri GG, Romao R, Yoshimura EM, Chammas MC. Low-level laser therapy in chronic autoimmune thyroiditis: a pilot study. Lasers Surg Med. 2010 Aug;42(6):589-96. doi: 10.1002/lsm.20941. PMID 20662037
- [Background] Hofling DB, Chavantes MC, Juliano AG, Cerri GG, Knobel M, Yoshimura EM, Chammas MC. Assessment of the effects of low-level laser therapy on the thyroid vascularization of patients with autoimmune hypothyroidism by color Doppler ultrasound. ISRN Endocrinol. 2012;2012:126720. doi: 10.5402/2012/126720. Epub 2012 Dec 17. PMID 23316383
- [Derived] Hofling DB, Chavantes MC, Buchpiguel CA, Cerri GG, Marui S, Carneiro PC, Chammas MC. Safety and Efficacy of Low-Level Laser Therapy in Autoimmune Thyroiditis: Long-Term Follow-Up Study. Int J Endocrinol. 2018 Nov 4;2018:8387530. doi: 10.1155/2018/8387530. eCollection 2018. PMID 30532779